CLINICAL TRIAL: NCT03801278
Title: An Expanded Access Study of Bemarituzumab (FPA144) for a Single Patient With Recurrent Bladder Cancer
Acronym: FPA144
Status: No longer available | Type: Expanded Access
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FPA144-006
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Recurrent Bladder Cancer
Keywords: Single patient
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — bemarituzumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: FPA144 — Bemarituzumab administration every two weeks
  Other Names: Bemarituzumab

SUMMARY:
This is an open-label, expanded access protocol to continue administration of bemarituzumab (FPA144) in a single patient with recurrent bladder cancer

DETAILED DESCRIPTION:
This protocol is intended to provide access to bemarituzumab (FPA144 an investigational agent) to a single patient with recurrent bladder cancer who had a response to study drug on FPA144-001. That study is closing and this expanded access protocol allows this single patient to continue receiving this agent.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign an Institutional Review Board-approved informed consent form prior to receiving bemarituzumab
2. Previously enrolled on the FPA144-001 study, received bemarituzumab and obtained clinical benefit from the investigational product (IP) administration

Exclusion Criteria:

1. Pregnancy and lactation

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult